CLINICAL TRIAL: NCT03046069
Title: FF/UMEC/VI: Qualitative Interviews and Discrete Choice Experiment(s) Evaluating the Perceived Benefits of the Features of FF/UMEC/VI (Single Inhaler Triple Therapy) Treatment in the UK, US and Germany
Brief Title: FF/UMEC/VI Inhaler: Qualitative Analysis and Subject Preference Survey
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: 206455
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Triple therapy; COPD; DCE; Qualitative
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Subjects included in telephone interviews: Approximately 10 subjects with COPD per country will be included in qualitative concept elicitation telephone interviews.
  Interventions: Other: Telephone interviews
- Subjects included in in-person focus groups: 1 in-person focus-group per country including up to 5 subjects with COPD will be included in the qualitative analysis.
  Interventions: Other: In-person focus groups
- Subjects included in DCE surveys- cognitive interviews: Up to six subjects with COPD in each of the UK, US and Germany will be asked to complete and provide feedback on the surveys.
  Interventions: Other: DCE surveys- cognitive interviews
- Subjects included in modified DCEs: Up to 20 subjects with COPD in each country will be included in pilot testing of the modified DCEs.
  Interventions: Other: Modified DCE
- Subjects included in Final DCE: 150 subjects with COPD in each of the UK, US and Germany will be included in the final online market specific DCE survey.
  Interventions: Other: Online DCE survey

INTERVENTIONS:
Other: Telephone interviews — Qualitative concept elicitation telephone interviews will be conducted in subjects with COPD to explore treatment effectiveness, symptoms, quality of life, and features of treatment that are considered to be most important to them when making treatment choices.
  Groups: Subjects included in telephone interviews
Other: In-person focus groups — Qualitative concept elicitation in-person focus groups will be conducted in subjects with COPD to explore treatment effectiveness, symptoms, quality of life, and features of treatment that are considered to be most important to them when making treatment choices.
  Groups: Subjects included in in-person focus groups
Other: DCE surveys- cognitive interviews — Draft version of the DCE surveys will be tested with subjects in cognitive interviews to explore the saliency of the attribute choices and assess whether the attributes are understandable, meaningful and comprehensive.
  Groups: Subjects included in DCE surveys- cognitive interviews
Other: Modified DCE — The modified DCEs will be piloted with subjects with COPD in each country to refine the underlying design and ensure that information is collected in an efficient way to enable the statistical analysis to be as precise as possible.
  Groups: Subjects included in modified DCEs
Other: Online DCE survey — An online DCE survey questionnaire will be given to the subjects to identify subject preferences, priorities and treatment goals.
  Groups: Subjects included in Final DCE

SUMMARY:
Three main classes of inhaled treatment exist for chronic obstructive pulmonary disease (COPD): Beta2-adrenergic agonists (which may be short (SABA) or long (LABA) acting), long-acting muscarinic acetylcholine receptor antagonists (LAMA), and inhaled corticosteroids (ICS). For subjects at higher risk of exacerbation, treatment with all these three classes of medication is recommended. This study aims to explore the potential utility of a device called single inhaler triple combination or fluticasone furoate/ umeclidinium/ vilanterol (FF/UMEC/VI) inhaler containing all three groups of compound. This is a mixed methods study with a qualitative phase and a quantitative Discrete Choice Experiment (DCE) phase and will be conducted in four stages: qualitative concept elicitation, DCE development, DCE piloting and testing, and conduct of the DCE. The study will conducted in the United Kingdom (UK), United States (US) and Germany and approximately 573 subjects with COPD will be included.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD, self-reported.
* Age: More than or equal to 40 years.
* Moderate to severe COPD, indicated by a COPD Assessment Test (CAT) score of greater than or equal to 10 or Modified Medical Research Council (MMRC) score of greater than or equal to 2.
* Currently prescribed and receiving one of the following treatment types: ICS/LABA; LABA/LAMA; ICS/LABA/LAMA (triple therapy); LAMA.
* Currently resident in the UK, US or Germany.
* Adequate written and oral fluency in language of country of residence.
* Willing and able to understand the study and provide informed consent.
* Has access to the internet (Cognitive interviews and DCE survey only).

Exclusion Criteria:

* Has taken part in any other stage of this study.
* Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD).
* Any co-morbidity that would inhibit the ability to provide informed consent or allow participation in a telephone of face-to-face interview.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with COPD who may be receiving any combination of dual or triple therapy treatment will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of the key relevant attributes of COPD treatment | Up to 368 hours
  The key attributes considered to be most important to subjects with COPD when making treatment choices will be assessed using the data from the subject interviews and focus groups.
Evaluation of the preferences, priorities and treatment goals of subjects with COPD for inhaled treatments | Up to 368 hours
  The probability of choosing one treatment over another will be evaluated using DCE survey questionnaire.

SECONDARY OUTCOMES:
Assessment of the relative appeal of different treatment approaches | Up to 371 hours
  The burden of COPD, priorities in terms of symptoms and treatment effect, goals and preferences of subjects will be analyzed.
Estimation of the relative importance of each attribute | Up to 371 hours
  The DCE online survey will be used to assess the relative importance of treatment attributes and priorities.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study 206455 can be found on the GSK Clinical Study Register. — https://www.gsk-studyregister.com/en/trial-details/?id=206455